CLINICAL TRIAL: NCT01681810
Title: An Open-Label Study of Oral Nitrite in Adults With Metabolic Syndrome and Hypertension
Brief Title: Oral Nitrite in Adults With Metabolic Syndrome and Hypertension
Acronym: ONTX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gladwin, Mark, MD (Individual)
Responsible Party: Principal Investigator, Kara S Hughan, MD, Assistant Professor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO11030131
Record Dates: First submitted 2012-07-03; First posted 2012-09-10 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Metabolic Syndrome; Hypertension
MeSH Terms: conditions — Metabolic Syndrome; Hypertension | interventions — Sodium Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14Nitrogen sodium nitrite (Experimental): sodium nitrite 40 mg three times a day for 12 weeks
  Interventions: Drug: 14Nitrogen Sodium Nitrite

INTERVENTIONS:
Drug: 14Nitrogen Sodium Nitrite — oral formulation of sodium nitrite 40 mg three times a day for 12 weeks
  Other Names: sodium nitrite

SUMMARY:
This research study is being conducted to examine the effects of daily inorganic nitrite treatment on the cardiometabolic and hormonal disturbances observed in overweight/obese adults with the metabolic syndrome and high blood pressure. Ultimately, oral nitrite therapy may have a major impact on the prevention and treatment of both diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
Cardiovascular disease remains the leading cause of death in the United States and worldwide. Several studies have demonstrated that fruit and vegetable rich diets significantly reduced blood pressure and reduced the risk of ischemic stroke and cardiovascular disease in general, the exact mechanisms remain poorly understood. Preclinical and clinical research over the last decade has revealed the important vasoprotective effects of nitrates and nitrites with regards to reduction in blood pressure, vascular inflammation and endothelial dysfunction. More recent findings suggest that inorganic nitrate and nitrite therapy may be involved in the regulation of glucose-insulin homeostasis.

For this reason, development of an oral formulation of nitrite salt represents a rational avenue of exploration for the treatment of cardiovascular diseases, whereby nitrite would ensure rapid acting effects upon absorption which can be further oxidized to nitrate via the enterosalivary circulation pathway. In this pathway, about 25% of circulating nitrate is concentrated in the saliva and reduced to nitrite by commensal mouth bacteria with nitrate reductase enzymes. The proposal is the first human study to investigate the inorganic nitrite effects (in any form) on insulin sensitivity in a patient population. This is the second human trial using orally delivered nitrite (previously as aqueous solution).

In the initial phase of the study, step up dosing and frequency of oral sodium nitrite to 40 mg three times daily occurred with no serious adverse events. After three subjects completed the study intervention on sodium nitrite 20 mg three times daily for 2 weeks followed by 40 mg three times daily for the remaining 10 weeks with no serious adverse events, all subjects in this current phase of the trial (n=20) began the 12-week study intervention with 40 mg three times daily. At the same time, in person monitoring visits (which included brief physical exams, directly observed nitrite dosing, secondary outcome measure assessment of methemoglobin level and blood pressure, interval histories, medication compliance review, symptom review and dispensing of study drug) were spaced from weekly intervals to subjects alternating weekly in person visits with phone visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Body mass index (BMI) greater than or equal to 30 kg/m^2
* Hypertension: defined as systolic blood pressure (SBP) greater than or equal to 130 and/or diastolic blood pressure (DBP) greater than or equal to 85 mm Hg
* Waist circumference: greater than 102 cm in men, greater than 88 cm in women

Exclusion Criteria:

* Positive urine pregnancy test or breastfeeding
* Concurrent use of medications affecting glucose metabolism (oral hypoglycemics, insulin, atypical antipsychotics)
* Recent addition or change in dosing of hormonal contraceptive medications [oral contraceptive pill (OCP), intrauterine device (IUD), DepoProvera]
* Current use of greater than or equal to 3 anti-hypertensive agents regardless of blood pressure control or normotensive on a single or double agent
* Current use of phosphodiesterase-5 inhibitors or organic nitrates
* Not stable on treatments for the prior three months or not planning to remain on current dose of medications for blood pressure, contraception, etc.
* Known chronic psychiatric or medical conditions including diabetes, liver or kidney disease or obesity syndromes
* Thyroid-stimulating hormone (TSH) greater than 8 milli-International unit/mL
* Smoker
* Anemia (central lab hemoglobin less than 11g/dL)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2018-02-08 (Actual); Study Completion 2018-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara S Hughan, MD, Principal Investigator — University of Pittsburgh; Mark Gladwin, MD, Study Director — University of Pittsburgh
Locations (1):
- Montefiore Hospital of University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Hughan KS, Levine A, Helbling N, Anthony S, DeLany JP, Stefanovic-Racic M, Goodpaster BH, Gladwin MT. Effects of Oral Sodium Nitrite on Blood Pressure, Insulin Sensitivity, and Intima-Media Arterial Thickening in Adults With Hypertension and Metabolic Syndrome. Hypertension. 2020 Sep;76(3):866-874. doi: 10.1161/HYPERTENSIONAHA.120.14930. Epub 2020 Aug 3. PMID 32755471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects 18-60 years with metabolic syndrome and hypertension were recruited through the University of Pittsburgh Research Participant Registry, University of Pittsburgh Nutrition and Obesity Research Center Registry, university and University of Pittsburgh Medical Center hospital electronic and paper advertising, and radio and bus advertising.
Pre-assignment Details: Twenty four age eligible subjects were consented and eligibility was confirmed. Four were excluded after eligibility confirmed due to poor IV access or not showing to baseline assessment visits, all prior to starting nitrite drug.
Period: Overall Study
Arm/Group | 14Nitrogen Sodium Nitrite
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants completing sodium nitrite 40 mg three times a day for 12 weeks
Arm/Group | 14Nitrogen Sodium Nitrite
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 52.4 [39 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Systolic blood pressure (SBP) [Mean (Standard Deviation); unit: mmHg] — Automated blood pressure was measured with a Dinamap DPC200X (GE Medical Systems Information Technology) after consent, history and physical examination. Subject was in the supine position with legs uncrossed and sitting upright in a chair in a quiet room.
  mmHg | 146 (15.7)
Diastolic blood pressure (DBP) [Mean (Standard Deviation); unit: mmHg] — Automated blood pressure was measured with a Dinamap DPC200X (GE Medical Systems Information Technology) after consent, history and physical examination. Subject was in the supine position with legs uncrossed and sitting upright in a chair in a quiet room.
  mmHg | 87.8 (8.57)
Mean arterial pressure (MAP) [Mean (Standard Deviation); unit: mmHg] — Automated blood pressure was measured with a Dinamap DPC200X (GE Medical Systems Information Technology) after consent, history and physical examination. Subject was in the supine position with legs uncrossed and sitting upright in a chair in a quiet room.
  mmHg | 109 (11.1)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Height and weight were measured in clothing without shoes. Height measured in centimeters (cm)by stadiometer and body weight measured in kilograms (kg) by Tanita scale. Measured height in cm converted to meters (m). BMI was calculated as weight (kg) divided by height (as m^2).
  kg/m^2 | 40.8 (6.63)
Waist circumference-male [Mean (Standard Deviation); unit: cm] — Measurement obtained in triplicate and 3 values averaged. Population: displaying sex-specific waist circumference as per eligibility criteria
  cm
    number analyzed (Participants) | 5
    (all) | 133.3 (11.82)
Waist circumference-female [Mean (Standard Deviation); unit: cm] — Measurement obtained in triplicate and 3 values averaged. Population: displaying sex-specific waist circumference as per eligibility criteria
  cm
    number analyzed (Participants) | 15
    (all) | 116.8 (13.07)
Thyroid stimulating hormone (TSH) [Mean (Standard Deviation); unit: mIU/mL] — TSH obtained by venipuncture.
  mIU/mL | 1.93 (1.45)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] — Hemoglobin obtained by venipuncture.
  g/dL | 14.1 (1.25)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Stimulated Glucose Disposal Over 12 Week Study Period
Description: Change in insulin stimulated glucose disposal was assessed during the 4-hour hyperinsulinemic euglycemic clamp at end of the 12 weeks and was compared to baseline (pre-nitrite). Insulin stimulated glucose disposal (mg/min) was calculated in the final 20 minutes of the 4-hour clamp at steady state and expressed as mg per kg lean body mass (as measured by DEXA) per minute. HumuLIN R regular insulin was infused at a rate of 40 microUnits/m2/min. A non-radioactive glucose isotope dilution (Isotec, Inc) was delivered as a primed, then constant infusion of the 98+% enriched stable isotope of D-glucose [6,6-D2] (0.22 umol x kg-1, 17.6 umol x kg-1 prime). Plasma glucose was clamped between 85-95 mg/dL with a variable infusion of 20% dextrose in water. The rate of dextrose infusion was adjusted based on arterialized plasma glucose measurements obtained every 5 minutes.
Time Frame: measured at 0 (baseline) and at 12 weeks
Population: The pre-drug hyperinsulinemic euglycemic clamp isotope data for 1 subject (used to determine insulin stimulated glucose disposal) was not interpretable despite repeat of the mass spectrometry assay. Therefore, the pre- and post- outcome measure for this subject was removed from analysis, giving a n=19 sample size for this analysis.
Measure: Mean (Standard Error); unit: mg/kg lean body mass/minute
Arm/Group | 14Nitrogen Sodium Nitrite
Number analyzed (Participants) | 19
mg/kg lean body mass/minute | 0.76 (0.58)
Statistical Analysis 1: Comparison: 14Nitrogen Sodium Nitrite; Test type: Other — Paired t-test comparing insulin stimulated glucose disposal at end of 12 weeks on nitrite drug to baseline (pre-drug) insulin stimulated glucose disposal; p = 0.2068, t-test, 2 sided

2. Secondary Outcome: Peak Change in Systolic Blood Pressure Over 12 Week Study Period
Description: Peak change in systolic blood pressure (SBP) on sodium nitrite compared to baseline. Subjects performed bi-weekly blinded automated blood pressures with a Dinamap DPC200X (GE Medical Systems Information Technology) in triplicate at study visits beginning 30 minutes after directly observed nitrite dosing. Five minute intervals were maintained between measurements while in the supine position with legs uncrossed and sitting upright in a hospital bed in a quiet room. The final 2 of 3 SBP measurements were averaged.
Time Frame: measured at 0 (baseline) and bi-weekly over 12 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | 14Nitrogen Sodium Nitrite
Number analyzed (Participants) | 20
mmHg | -10.45 (3.01)
Statistical Analysis 1: Comparison: 14Nitrogen Sodium Nitrite; Test type: Other — One-way repeated measures ANOVA comparing blood pressure over time on nitrite drug to baseline (pre-drug) blood pressure; p = 0.0074, ANOVA — Bonferroni adjusted p-value for multiple comparisons

3. Secondary Outcome: Peak Change in Diastolic Blood Pressure Over 12 Week Study Period
Description: Peak change in diastolic blood pressure (DBP) on sodium nitrite compared to baseline. Subjects performed bi-weekly blinded automated blood pressures with a Dinamap DPC200X (GE Medical Systems Information Technology) in triplicate at study visits beginning 30 minutes after directly observed nitrite dosing. Five minute intervals were maintained between measurements while in the supine position with legs uncrossed and sitting upright in a hospital bed in a quiet room. The final 2 of 3 DBP measurements were averaged.
Time Frame: measured at 0 (baseline) and bi-weekly over 12 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | 14Nitrogen Sodium Nitrite
Number analyzed (Participants) | 20
mmHg | -13.05 (2.2)
Statistical Analysis 1: Comparison: 14Nitrogen Sodium Nitrite; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANOVA — Bonferroni adjusted p-value for multiple comparisons

4. Secondary Outcome: Peak Change in Mean Arterial Pressure Over 12 Week Study Period
Description: Peak change in mean arterial pressure (MAP) on sodium nitrite compared to baseline. Subjects performed bi-weekly blinded automated blood pressures with a Dinamap DPC200X (GE Medical Systems Information Technology) in triplicate at study visits beginning 30 minutes after directly observed nitrite dosing. Five minute intervals were maintained between measurements while in the supine position with legs uncrossed and sitting upright in a hospital bed in a quiet room. The final 2 of 3 MAP measurements were averaged.
Time Frame: measured at 0 (baseline) and bi-weekly over 12 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | 14Nitrogen Sodium Nitrite
Number analyzed (Participants) | 20
mmHg | -12.00 (2.15)
Statistical Analysis 1: Comparison: 14Nitrogen Sodium Nitrite; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANOVA — Bonferroni adjusted p-value for multiple comparisons

5. Secondary Outcome: Peak Change in Methemoglobin Over 12 Week Study Period
Description: Peak change in methemoglobin on sodium nitrite compared to baseline. Methemoglobin was assessed bi-weekly at study visits 30 minutes after directly observed nitrite dosing using noninvasive co-oximetry (Masimo Corp, Irvine, CA).
Time Frame: measured at 0 (baseline) and bi-weekly over 12 weeks
Measure: Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | 14Nitrogen Sodium Nitrite
Number analyzed (Participants) | 20
percentage of total hemoglobin | 0.42 (0.11)
Statistical Analysis 1: Comparison: 14Nitrogen Sodium Nitrite; Test type: Other — One-way repeated measures ANOVA comparing methemoglobin percent over time on nitrite drug to baseline (pre-drug) methemoglobin percent; p = 0.0127, ANOVA — Bonferroni adjusted p-value for multiple comparisons

ADVERSE EVENTS:
Time Frame: Adverse event (AE) collection occurred throughout 12 weeks of study drug treatment until 1 month after completing study drug.
Description: Adverse event (AE) collection occurred after eligibility was confirmed. AE collection was then queried bi-weekly by standard questionnaire, daily by standard diary card logged by participants, and with regular investigator assessment. First AE assessment began at first baseline assessment study visit prior to first dose of study drug visit.
Arm/Group | 14Nitrogen Sodium Nitrite
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 14Nitrogen Sodium Nitrite (N=20)
Abdominal pain (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 15 (62)
Dizziness (Nervous system disorders) | 5 (14)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (10)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Flushing (Vascular disorders) | 5 (5)
Tachycardia (Cardiac disorders) | 2 (5)
Fatigue (General disorders) | 2 (3)
Upper respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 9 (15)
Dry mouth (Skin and subcutaneous tissue disorders) | 6 (15)
Sore mouth (Skin and subcutaneous tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (21)
Joint pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Arm/hand pain (non-joint) (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgias (Musculoskeletal and connective tissue disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (5)
Sleep disruption (General disorders) | 2 (9)

LIMITATIONS AND CAVEATS:
The pre-drug clamp isotope data for 1 subject (used to determine insulin stimulated glucose disposal) was uninterpretable, despite repeating the mass spectrometry assay. Subject's isotope data was removed from analysis (n=19 analysis sample size).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT01681810/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT01681810/ICF_001.pdf